CLINICAL TRIAL: NCT01735110
Title: A Prospective, Multicenter, Randomized Trial Assessing the Safety and Efficacy of PCI Via Radial Versus Femoral Approach in Patients With Left Main and/or Three-Vessel Disease
Brief Title: PREPARE：Assessing the Safety and Efficacy of Radial Versus Femoral Approach PCI
Acronym: PREPARE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Medtronic (Industry); CCRF Consulting Co., Ltd. (Other)
Responsible Party: Principal Investigator, Yuejing Yang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREPARE
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Transradial-transfemoral Coronary Interventions Comparison

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoral approach group (Active Comparator): PCI through Femoral approach
  Interventions: Procedure: transfemoral intervention (TFI)
- radial approach group (Experimental): PCI through radial approach
  Interventions: Procedure: Transradial intervention

INTERVENTIONS:
Procedure: transfemoral intervention (TFI)
  Arms: Femoral approach group
Procedure: Transradial intervention
  Arms: radial approach group

SUMMARY:
The purpose of PREPARE trial is to evaluate the long-term safety and efficacy of TRI versus TFI for PCI in patients with left main (LM) and/or three-vessel coronary artery disease.

DETAILED DESCRIPTION:
Transradial intervention (TRI) has been widely practiced in China, accounting for approximate 80 to 90% of procedures. A recent meta-analysis indicated that TRI has advantages in reducing major bleeding and ischemic events compared to transfemoral intervention (TFI) after the percutaneous coronary intervention (PCI). However, no clinical trial has yet shown statistical equivalence in terms of long-term efficacy of TRI compared with TFI for the treatment of complex coronary lesions, which is simply due to limited numbers of subjects enrolled. The purpose of PREPARE trial is to evaluate the long-term safety and efficacy of TRI versus TFI for PCI in patients with left main (LM) and/or three-vessel coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age.
* Patient is able to verbally acknowledge an understanding of the associated risks, benefits and treatment alternatives and he or his legally authorized representative provides written informed consent prior to the randomization, as approved by the appropriate IEC.
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible changes in the electrocardiogram (ECG) consistent with ischemia).
* Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
* Patient with complex lesion who may need two or more than 2 stents implantation during the indexed procedure is required surgeon's consultation before the operation. The surgical consultation outcome must be recorded in detail.
* Patient must agree to undergo all protocol-required follow-up examinations.
* Patient must agree not to participate in any other clinical study within the duration of this trial.

Angiographic inclusion criteria：

* Target lesion must be able to be treated by using six-French guiding catheters.
* Target lesion can be Left Main and/or Multivessel Diseases with Syntax score ≤32 for LM and Syntax score ≤22 for MVD.

Exclusion Criteria:

* Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant.
* Patient is receiving or scheduled to receive chemotherapy for malignancy.
* Patient is receiving immunosuppression therapy or has known immunosuppressive or autoimmune disease (e.g. Human Immunodeficiency Virus, Lupus etc. Not include diabetes mellitus).
* Known hypersensitivity or contraindication to aspirin, zotarolimus, polymer, Nickel, cobalt, chromium, iron, tungsten, etc. or stainless steel.
* Patient has extensive peripheral vascular disease that precludes safely insertion of 6 French sheath.
* Patient has other medical illness (e.g., cancer or congestive heart failure) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
* Female patients of childbearing potential who have refused a urine or blood pregnancy test (to be done within 7 days prior to index procedure), patients who are nursing at the time of index procedure and those patients who do not agree at the time of consent to use any approved form of birth control up to and including the follow-up at 1 year.
* STEMI within 72h prior to procedure.
* History of CABG.
* Radial artery or femoral artery presence serious vascular bend or deformity that the 6F sheath can not go though.
* Based on investigator's clinical judgments, high-risk patients, referring to predicted procedural risks being higher than the procedural benefits must be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiac and cerebrovascular events (MACCE) at 12 months | 1 year
  The primary endpoint is the major adverse cardiac and cerebrovascular events (MACCE) defined as the composite of all-caused death, all stroke, all myocardial infarction (MI), or any revascularization at 12 months.

SECONDARY OUTCOMES:
The second endpoint is the rate of first occurrence of bleeding complication (BARC Definition type 3 and 5) at 7 days post-procedure | 7 days
  - The second endpoint is the rate of first occurrence of bleeding complication (BARC Definition type 3 and 5) at 7 days post-procedure

OTHER OUTCOMES:
Other outcomes | 5years
  * Death (Cardiac, Vascular, Non-cardiovascular)
  * MI
  * Stroke
  * TLR (Ischemia-driven, not ischemia-driven) at 12 months
  * TVR (Ischemia-driven, not ischemia-driven) at 12 months
  * Stent thrombosis (per ARC definition) at 12 months
  * Minor bleeding complication (BARC type 1 or 2) at 7 and 30 days
  * Total bleeding complication (BARC definition) at 7 and 30 days
  * PCI procedural success
  * Device success
  * Procedural or fluoro time
  * Cross lesion failure rate
  * Total procedure time
  * Total amount of contrast use
  * Total radiation doses
  * Major vascular access site complication at discharge and 30 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yuejing Yang, Professor, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital